CLINICAL TRIAL: NCT05784168
Title: The Effect of Manual Therapy and Therapeutic Exercises on Pain and Functional Status in Persons With Chronic Non-specific Low Back Pain
Brief Title: The Effect of Manual Therapy and Therapeutic Exercises on Pain and Functional Status in Persons With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LithuanianSportsU12
Record Dates: First submitted 2023-02-24; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
Keywords: low back pain; manual therapy; exercise therapy
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (Experimental): 6 weeks, 12 sessions in total, 2 times a week of manual therapy: spinal manipulation, specific mobilisations and stretches. Manual therapy treatments are carried out by a physiotherapist with more than 10 years of experience.
  In addition, 6 weeks, 5 times a week, a programme of therapeutic exercises at home: muscle strengthening and stretching, balance and coordination training, spinal stabilisation exercises.
  Interventions: Other: Manual therapy
- Exercise therapy (Experimental): 6 weeks, 12 sessions in total, 2 times a week therapeutic exercise programme under the supervision of a physiotherapist. The exercise programme consisted of muscle strengthening and stretching, balance and coordination training, spinal stabilisation exercises.
  In addition, 6 weeks, 5 times a week, a programme of therapeutic exercises at home: muscle strengthening and stretching, balance and coordination training, spinal stabilisation exercises.
  Interventions: Other: Exercise therapy

INTERVENTIONS:
Other: Manual therapy — 6 weeks, 12 sessions in total, 2 times a week of manual therapy: spinal manipulation, specific mobilisations and stretches. Manual therapy treatments are carried out by a physiotherapist with more than 10 years of experience.
  In addition, 6 weeks, 5 times a week, a programme of therapeutic exercises at home: muscle strengthening and stretching, balance and coordination training, spinal stabilisation exercises.
  Arms: Manual therapy
Other: Exercise therapy — 6 weeks, 12 sessions in total, 2 times a week therapeutic exercise programme under the supervision of a physiotherapist. The exercise programme consisted of muscle strengthening and stretching, balance and coordination training, spinal stabilisation exercises.
  In addition, 6 weeks, 5 times a week, a programme of therapeutic exercises at home: muscle strengthening and stretching, balance and coordination training, spinal stabilisation exercises.
  Arms: Exercise therapy

SUMMARY:
Non-specific chronic low back pain (LBP) can be managed with a variety of treatments such as educational programmes, behavioural therapy, acupuncture, medication, electrophysical agents, manual therapy and exercise therapy. Although the above therapies are widely used, they show limited effect at best, with frequent recurrences of LBP. There is insufficient data to prove that one type of exercise is superior to another. Manual therapy is a common therapeutic method used in the treatment of LBP. Therefore, we hypothesised that manual therapy combined with therapeutic exercises would lead to a greater reduction in back pain and improvement in functional status. The aim of the study was to evaluate the effect of 6 weeks of manual therapy combined with therapeutic exercise on pain and functional status in subjects with chronic non-specific low back pain.

DETAILED DESCRIPTION:
The individuals with chronic non-specific low back pain participated in the study. Subjects were randomly divided into two groups: physiotherapy and manual therapy. All the participants received 12 intervention sessions. In addition, all subjects exercised at home 5 days a week. Subjects' back static strength endurance was assessed by the ITO test, abdominal muscle static strength endurance was assessed by the Kraus-Webber test, fear of movement by the TAMPA kinesiophobia test, torso mobility by the Schober test, pain by the numerical analogy scale. Functional status was assessed by Oswestry and Roland-Morris questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain (>8 weeks);
* Persons of working age;
* Must be able to perform therapeutic exercises.

Exclusion Criteria:

* Severe cardiovascular disease;
* Oncological disorders;
* Neurological symptoms of disorders;
* Osteoarthritis;
* Spondylolisthesis and spondylosis;
* Radiculopathy;
* Myelopathy;
* Spinal fracture.
* Pregnancy or lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain at 6 weeks | Baseline and after 6 weeks
  Pain was assessed using a Numerical Rating Scale (NRS) that used a 10-cm line with end-point descriptors such as 'no pain' marked at the left end and 'worst pain imaginable' marked at the right end. Patients were asked to mark a point on the line that best represented their pain at the time of the evaluation. The distance from 'no pain' to the patient's mark was then measured and recorded as the NRS score: 0 cm was defined as no pain, 1-3 cm as mild pain, 4 or 5 cm as moderate pain, 6-8 cm as severe pain and 9 or 10 cm as the worst pain imaginable.
Change from baseline Oswestry Disability Index for functional status at 6 weeks | Baseline and after 6 weeks
  The Oswestry questionnaire (ODI) was used to assess the impact of back pain on functional status and disability. It consists of ten questions (pain intensity, self-care, lifting objects, walking, sitting, standing, sleeping, sexual life, social life and travelling). There are six answer options for each question, and the value of each question ranges from 0 (no problems/no disability) to 5 (major problems/major disability in this area). The total ODI score is calculated as the sum of the scores for each question and the total ODI score ranges from 0 to 50. The percentage of scores is calculated as follows: sum of scores / 50 x 100 = percentage (%). The lower the score, the lower the impact of pain on functional status.
Change from baseline Roland Morris Disability Questionnaire at 6 weeks | Baseline and after 6 weeks
  The Roland Morris Disability Questionnaire consists of 24 statements relating to daily living and physical activities such as personal care, sleep, work and walking. The scale ranges from 0 to 24, with the highest score indicating maximum functional disability.
Change from baseline Mobility of the lumbar spine at 6 weeks | Baseline and after 6 weeks
  The Schober test was used to assess lumbar spine mobility. The test is performed with the subject standing upright, arms at the sides, and the examiner locates the midline between the iliac crests, on the dorsal side, and marks the first point there. A second point is marked 10 cm above the first point. 5 cm below the first marked point, a third point shall be marked. The subject is then asked to bend forward as far as he or she can without pain and without bending the knees, and the distance between the first and the third point is measured with a centimetre tape. The test is negative if the distance between the marked points is 7 cm or more and positive if the distance is less than 7 cm, indicating limited mobility of the lumbar spine.
Change from baseline Abdominal muscle static endurance at 6 weeks | Baseline and after 6 weeks
  Static abdominal muscle endurance test - Kraus-Weber. The subject lies on the back, knees bent at 90 degrees, arms crossed over the chest. The subject flexes the thorax, i.e. pulls the lower shoulder blade away from the surface, and is isometrically holds the body in this position. The test is terminated if the subject remains in this position for more than 300 seconds. The test shall be terminated when the lower scapular angle descends downwards and is no longer maintained or when the subject experiences unpleasant sensations and/or pain.
Change from baseline Back muscle static endurance at 6 weeks | Baseline and after 6 weeks
  Static back muscle endurance test - Ito. The subject lies on his/her stomach, arms at his/her sides, palms up. The subject lifts the upper trunk to the lower sternum from the lying surface. The test is terminated if the subject remains standing for more than 300 seconds. If the subject does not maintain the position and touches the ground or experiences unpleasant sensations and/or pain, the test shall also be terminated.
Change from baseline Kinesiophobia at 6 weeks | Baseline and after 6 weeks
  The Tampa Scale of Kinesiophobia was used to assess the fear of movement or repetitive trauma in pain patients. The highest score indicates a high level of kinesiphobia.

CONTACTS AND LOCATIONS:
Overall Officials: Vytautas Pilelis, Master, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No